CLINICAL TRIAL: NCT02753946
Title: Randomized, Double-Blind, Comparative Study to Evaluate the Safety and Efficacy of ZTI-01 vs Piperacillin/Tazobactam in the Treatment of cUTI/AP Infection in Hospitalized Adults
Brief Title: Safety and Efficacy of ZTI-01 (IV Fosfomycin) vs Piperacillin/Tazobactam for Treatment cUTI/AP Infections
Acronym: ZEUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nabriva Therapeutics AG (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZTI-01-200; 2015-003372-73 (EudraCT Number)
Record Dates: First submitted 2016-04-13; First posted 2016-04-28 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Urinary Tract Infection Symptomatic; Acute Pyelonephritis; Urinary Tract Infection Complicated
MeSH Terms: interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZTI-01 (Experimental): 6 g ZTI-01 (IV fosfomycin) intravenously administered every 8 hours (18g total daily dose for 7-14 calendar days)
  Interventions: Drug: ZTI-01
- piperacillin tazobactam (Active Comparator): 4.5 g piperacillin/tazobactam (4 g piperacillin/0.5 g tazobactam) intravenously administered every 8 hours (13.5g total daily dose for 7-14 calendar days)
  Interventions: Drug: Piperacillin-tazobactam

INTERVENTIONS:
Drug: ZTI-01 — 6g ZTI-01 intravenous infusion TID q8 hours
  Other Names: disodium fosfomycin
  Arms: ZTI-01
Drug: Piperacillin-tazobactam — 4.5g piperacillin-tazobactam intravenous infusion TID q8 hours
  Other Names: piperacillin-tazobactam combination product
  Arms: piperacillin tazobactam

SUMMARY:
The purpose of the study is to demonstrate the safety and efficacy of ZTI-01 (IV fosfomycin) as non-inferior to piperacillin/tazobactam in overall success (clinical cure and microbiologic eradication) for the treatment of hospitalized patients with complicated urinary tract infections (cUTI) or acute pyelonephritis (AP).

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel-group study to evaluate the safety, tolerability, efficacy, and pharmacokinetics of ZTI-01 (IV fosfomycin) compared to piperacillin/tazobactam in the treatment of hospitalized adults with cUTI or AP. Diagnosed and prescreened hospitalized patients will be randomized 1:1 to receive one of two intravenous treatments: 6 g ZTI-01 three times daily (18g total daily dose) or 4.5 g piperacillin/tazobactam three times daily (13.5g total daily dose) for 7 calendar days, with option to extend treatment up to 14 days in patients with positive blood culture at pretreatment. Patients will participate in the study for approximately 26 days. Urine cultures will be obtained and organisms quantified for qualified patients at baseline, during treatment, at end of treatment (EOT), at test of cure (TOC) and late follow up visits (LFU). Blood cultures will be obtained at baseline and repeated if positive throughout the study. Safety and efficacy evaluations will include vital signs, labs, physical exams, ECG and overall response as evaluated by the Investigator. Pharmacokinetic samples will be obtained (sparse sampling) for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent form (ICF);
2. Male or female, at least 18 years of age;
3. Diagnosis requires hospitalization and treatment with intravenous (IV) antibiotics;
4. Documented or suspected cUTI or AP including at least 2 protocol defined signs and symptoms and a urine specimen with evidence of pyuria plus at least one protocol defined associated risk
5. Pretreatment baseline urine culture specimen
6. Expectation that any implanted urinary instrumentation will be removed or replaced not longer than 24 hours, after randomization;
7. Expectation that patient will survive anticipated duration of the study;
8. Patient requires initial hospitalization to manage the cUTI or AP;
9. Women of childbearing potential have had a negative pregnancy test before randomization and be willing to consistently use a highly effective method of contraception
10. Male study participants will be required to use condoms with a spermicide throughout study

Exclusion Criteria:

1. Presence of any of the following conditions: perinephric abscess, renal corticomedullary abscess, uncomplicated urinary tract infection, recent history of trauma to the pelvis or urinary tract, polycystic kidney disease, chronic vesicoureteral reflux, previous or planned renal transplantation; patients receiving dialysis/hemodialysis/CVVH, previous or planned cystectomy or ileal loop surgery; known or suspected infection; caused by pathogen resistant to study treatment antibiotics
2. Presence of suspected or confirmed acute bacterial prostatitis, orchitis, epididymitis, or chronic bacterial prostatitis as determined by history and/or physical examination;
3. Gross hematuria requiring intervention;
4. Urinary tract surgery within 7 days prior to randomization or urinary tract surgery planned during the study period;
5. Creatinine clearance <20 mL/min using the Cockcroft-Gault formula;
6. Non-renal source of infection such as endocarditis, osteomyelitis, abscess, meningitis, or pneumonia diagnosed within 7 days prior to randomization;
7. Signs of severe sepsis as defined per protocol;
8. Pregnant or breastfeeding women;
9. Known seizure disorder requiring current treatment with anti-seizure medication which would prohibit the patient from complying with the protocol;
10. Cancer chemotherapy, immunosuppressive medications for transplantation, or medications for rejection of transplantation with 30 days of randomization;
11. Significant hepatic disease or dysfunction, including known acute viral hepatitis or hepatic encephalopathy;
12. ALT/AST >5 × ULN or total bilirubin >3 × ULN at Screening;
13. Receipt of any potentially-effective systemic antibiotic with activity against Gram-negative uropathogens for more than 24 hours within the 72-hour window prior to randomization (exceptions defined in protocol);
14. Requirement for additional systemic antibiotic therapy (other than study drug) or antifungal therapy for vaginal candidiasis;
15. Likely to require the use of an antibiotic for cUTI or AP prophylaxis during the study;
16. Known history of HIV virus infection and known recent CD4 count <200/mm3;
17. Presence of significant immunodeficiency or an immunocompromised condition and long-term use of systemic corticosteroids;
18. Presence of neutropenia;
19. Presence of thrombocytopenia;
20. A QT interval corrected using Fridericia's formula >480 msec;
21. History of significant hypersensitivity or allergic reaction to fosfomycin, any contraindication to the use of piperacillin/tazobactam;
22. Participation in a clinical study involving investigational medication or investigational device within the last 30 days prior to randomization;
23. Inability, in the judgment of the Investigator, to tolerate the salt load required for study drug administration;
24. Unable or unwilling, in the judgment of the Investigator, to comply with the protocol;
25. Any patients previously randomized in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn J Ellis-Grosse, PhD, Study Chair — Zavante Therapeutics, Inc.
Locations (68):
- United States (6):
  - Pensacola, Florida
  - Augusta, Georgia
  - Columbus, Georgia
  - Boylston, Massachusetts
  - St Louis, Missouri
  - Butte, Montana
- Belarus (5):
  - Brest
  - Grodno
  - Homyel
  - Minsk
  - Vitebsk
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Croatia (3):
  - Slavonski Brod
  - Split
  - Zagreb
- Czechia (3):
  - Brno
  - Hradec Králové
  - Liberec
- Estonia (2):
  - Kohtla-Järve
  - Tallinn
- Georgia (3):
  - Batumi
  - Kutaisi
  - Tbilisi
- Greece (3):
  - Ampelokipoi
  - Athens
  - Thessaloniki
- Hungary (6):
  - Budapest
  - Miskolc
  - Nagykanizsa
  - Pécs
  - Szekszárd
  - Szentes
- Latvia (2):
  - Riga
  - Valmiera
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (7):
  - Bielsko-Biala
  - Krakow
  - Lodz
  - Piaseczno
  - Tychy
  - Wroclaw
  - Zamość
- Romania (3):
  - Bucharest
  - Craiova
  - Oradea
- Russia (11):
  - Krasnoyarsk
  - Moscow
  - Moscow, Zelenograd
  - Nizhny Novgorod
  - Novosibirsk
  - Penza
  - Rostov-on-Don
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Vsevolozhsk
- Slovakia (3):
  - Martin
  - Poprad
  - Žilina
- Ukraine (6):
  - Chernihiv
  - Dnipropetrovsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Yes
Individual IPD data will be shared in listings with FDA, IRB/ECs, Data Monitoring Committee
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: ongoing submissions to IND
Access Criteria: IND/NDA submission, CTA submissions

REFERENCES:
- [Derived] Kaye KS, Rice LB, Dane AL, Stus V, Sagan O, Fedosiuk E, Das AF, Skarinsky D, Eckburg PB, Ellis-Grosse EJ. Fosfomycin for Injection (ZTI-01) Versus Piperacillin-tazobactam for the Treatment of Complicated Urinary Tract Infection Including Acute Pyelonephritis: ZEUS, A Phase 2/3 Randomized Trial. Clin Infect Dis. 2019 Nov 27;69(12):2045-2056. doi: 10.1093/cid/ciz181. PMID 30861061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with cUTI/AP based on signs and symtoms requiring 7 days hospitalization (or up to 14 days in case of bacteremia). No oral switch is allowed in the study.
  Confirmatory microbiology data only available after randomization.
Pre-assignment Details: At least 30% of patients required a diagnosis of AP. Receipt of effective systemic antibiotic for >24 hrs within 72-hr window before randomization exclusionary but receiving single dose of short-acting systemic antibiotic within 72 hrs of randomization permitted up to a max of 25% of the study enrollments.
Period: Overall Study
Arm/Group | ZTI-01 | Piperacillin Tazobactam
Started (465 were randomized but 1 randomized patient had adverse event prior to dosing) | 233 | 231
Completed | 219 | 222
Not Completed | 14 | 9
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: All subjects included (note 1 subject randomized discontinued prior to dosing). Note 6 subjects were incorrectly identified as Hispanic or Latino, instead of White in the database; errata recorded to file.
Groups:
- Total: Total of all reporting groups
Arm/Group | ZTI-01 | Piperacillin Tazobactam | Total
Number analyzed (Participants) | 233 | 232 | 465
Age, Customized [Count of Participants; unit: Participants]
  < 65 years of age | 159 | 155 | 314
  65 to 75 years of age | 52 | 42 | 94
  > 75 years of age | 22 | 35 | 57
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 146 | 297
  Male | 82 | 86 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 233 | 232 | 465
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 233 | 232 | 465
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 6 | 2 | 8
  Hungary | 4 | 5 | 9
  United States | 1 | 0 | 1
  Czechia | 7 | 7 | 14
  Ukraine | 71 | 73 | 144
  Belarus | 39 | 31 | 70
  Russia | 39 | 39 | 78
  Latvia | 13 | 16 | 29
  Poland | 10 | 12 | 22
  Georgia | 11 | 14 | 25
  Slovakia | 8 | 16 | 24
  Bulgaria | 6 | 4 | 10
  Lithuania | 6 | 7 | 13
  Croatia | 5 | 3 | 8
  Estonia | 7 | 3 | 10
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m2] — Population: 1 subject randomized discontinued prior to treatment
  kg/m2
    number analyzed (Participants) | 233 | 231 | 464
    (all) | 25.81 (5.355) | 26.44 (6.167) | 26.12 (5.776)
Screening Creatinine Clearance Group [Count of Participants; unit: Participants] — Cockroft Gault Equation used Population: Note 1 subject randomized discontinued prior to treatment due to an adverse event
  Participants
    <20 mL/min: number analyzed (Participants) | 232 | 232 | 464
    <20 mL/min | 0 | 0 | 0
    > or = 20 to 30 mL/min: number analyzed (Participants) | 232 | 232 | 464
    > or = 20 to 30 mL/min | 4 | 1 | 5
    >30 to 40 mL/min: number analyzed (Participants) | 232 | 232 | 464
    >30 to 40 mL/min | 12 | 7 | 19
    >40 to 50 mL/min: number analyzed (Participants) | 232 | 232 | 464
    >40 to 50 mL/min | 16 | 19 | 35
    > 50 mL/min: number analyzed (Participants) | 232 | 232 | 464
    > 50 mL/min | 200 | 205 | 405

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Overall Success
Description: Clinical cure (resolution or significant improvement in signs and symptoms) and microbiologic eradication (baseline pathogen) in m-MITT population
Time Frame: TOC Visit (Day 19)
Population: Microbiologic Modified Intent-to-Treat (m-MITT) population was used to assess overall success.
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 | Piperacillin Tazobactam
Number analyzed (Participants) | 184 | 178
Participants | 119 | 97

2. Secondary Outcome: Number of Patients With a Response of Clinical Cure in Various Protocol Populations
Description: mMITT
Time Frame: TOC Visit (Day 19)
Population: Microbiologic Modified Intent-to-Treat (m-MITT) population was used to assess clinical cure.
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 | Piperacillin Tazobactam
Number analyzed (Participants) | 184 | 178
Participants | 167 | 163

3. Secondary Outcome: Number of Patients With a Response of Microbiologic Eradication
Description: mMITT
Time Frame: TOC Visit (Day 19)
Population: Microbiologic Modified Intent-to-Treat (m-MITT) population was used to assess microbiologic eradication.
Measure: Count of Participants; unit: Participants
Arm/Group | ZTI-01 | Piperacillin Tazobactam
Number analyzed (Participants) | 184 | 178
Participants | 121 | 100

ADVERSE EVENTS:
Arm/Group | ZTI-01 | Piperacillin Tazobactam
All-Cause Mortality (participants affected / at risk) | 0/233 | 0/231
Serious Adverse Events (participants affected / at risk) | 5/233 | 6/231
Other Adverse Events (participants affected / at risk) | 55/233 | 31/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZTI-01 (N=233) | Piperacillin Tazobactam (N=231)
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1
Acute Media Otitis (Infections and infestations) | 1 | 0
Prostatic Abscess (Infections and infestations) | 1 | 0
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Abscess (Infections and infestations) | 0 | 1
Septic Embolus (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZTI-01 (N=233) | Piperacillin Tazobactam (N=231)
Nausea (Gastrointestinal disorders) | 10 | 3
Diarrhea (Gastrointestinal disorders) | 9 | 11
Vomiting (Gastrointestinal disorders) | 9 | 1
Infusion site phlebitis (General disorders) | 2 | 6
Alanine aminotransferase increased (Investigations) | 20 | 6
Aspartate aminotransferase increased (Investigations) | 17 | 6
Hypokalemia (Metabolism and nutrition disorders) | 14 | 3
Headache (Nervous system disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days